CLINICAL TRIAL: NCT01287390
Title: Adaptive, Image-guided, Intensity-modulated Radiotherapy for Head and Neck Cancer in the Reduced Volumes of Elective Neck: a Multicenter, Two-arm, Randomized Phase II Trial.
Brief Title: Adaptive, Image-guided, Intensity-modulated Radiotherapy for Head and Neck Cancer in the Reduced Volumes of Elective Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/012
Record Dates: First submitted 2011-01-26; First posted 2011-02-01 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Primary Non-operated Squamous Cell Carcinoma of Oral Cavity; Primary Non-operated Squamous Cell Carcinoma of Oropharynx; Primary Non-operated Squamous Cell Carcinoma of Hypopharynx; Primary Non-operated Squamous Cell Carcinoma of Larynx
Keywords: squamous cell carcinoma; oral cavity; oropharynx; hypopharynx; larynx
MeSH Terms: conditions — Carcinoma, Squamous Cell; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard radiotherapy treatment (Active Comparator): These patients receive the normal standard treatment.
  Interventions: Procedure: video fluoroscopy; Other: scoring acute toxicity; Other: scoring of late toxicity; Other: scoring quality of life (QOL)
- adaptive radiotherapy (Experimental): These patients receive the adaptive image-guided intensity-modulated radiotherapy (IMRT) for head and neck cancer.
  Interventions: Procedure: video fluoroscopy; Procedure: extra imaging; Other: scoring acute toxicity; Other: scoring of late toxicity; Other: scoring quality of life (QOL)

INTERVENTIONS:
Procedure: video fluoroscopy — video fluoroscopy of swallowing function at baseline, 6 months and 12 months follow-up
Procedure: extra imaging — For tumor response, 2 extra CT or Fludeoxyglucose (18F)-Positron Emission Tomography (PET)/Computed Tomography (CT), and/or Magnetic Resonance Imaging (MRI) will be performed.
  Arms: adaptive radiotherapy
Other: scoring acute toxicity — Acute toxicity scoring, based on Common Toxicity criteria (CTC) version 2.
Other: scoring of late toxicity — Scoring of late toxicity with the 'late effects in normal tissues subjective, objective, management and analytic'(LENT-SOMA) scale.
Other: scoring quality of life (QOL) — Quality of life is scored with the Quality of Life Questionnaire of the 'European Organisation for Research and Treatment of Cancer' (EORTC QOL-C30) and the Head and Neck Cancer Specific Quality of Life Questionnaire (QLQ-H&N 35).

SUMMARY:
Severe acute and late dysphagia is now considered as a dose-limiting toxicity of radio(chemo)therapy for head and neck cancer that significantly affects patients' quality of life. We propose to preserve swallowing function by:

* adapting (individualizing) treatment (intensity-modulated radiotherapy: IMRT) to per-treatment changes occurring in the tumor and surrounding organs and tissues;
* reducing the volumes of elective neck, that may result in significant decrease of severe acute and late dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx and larynx.
* Primary non-resected tumor and/or patients refused surgery
* Stage T1-4, N0-3; for cancer of the glottis T3-4 or T any N1-3
* Decision of curative radiotherapy or radiochemotherapy made by a Multidisciplinary Group of Head and Neck Tumors at UZ Gent and UZ Gasthuisberg Leuven
* Karnofsky performance status >= 70 %
* Age >= 18 years old
* Informed consent obtained, signed and dated before specific protocol procedures

Exclusion Criteria:

* Treatment combined with brachytherapy
* Prior irradiation to the head and neck region
* Surgery of the primary tumor except lymph node dissection prior to radiotherapy
* induction chemotherapy
* history of prior malignancies, except for cured non-melanoma skin cancer, curatively treated in-situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease at least 5 years
* Distant metastases
* Creatinine clearance (Cockroft-Gault) =< 60 milliliter/minute before treatment or creatinine value > 1,3 milligram/deciliter
* Known allergy to the CT-contrast agents
* Pregnant or lactating women
* Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study
* Patient unlikely to comply with protocol, i.e. uncooperative attitude, inability to return for follow-up visits and unlikely to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Reduction of acute and late treatment-induced dysphagia | after 1 year
  Reduction of the rates of acute and late treatment-induced dysphagia with experimental treatment as compared to standard treatment.

SECONDARY OUTCOMES:
acute treatment-induced toxicity | weekly during treatment
late treatment-induced toxicity | after 1, 3, 6, 9 and 12 months
tumor response: imaging | after 3 months
tumor response: clinical examination | after 1, 3, 6, 9 and 12 months
local, regional and distant control: imaging | after 3 months
local, regional and distant control: clinical examination | after 1,3, 6, 9 and 12 months
local, regional and distant control: biopsy | from 3 months on

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, PhD, MD, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - University Hospital Ghent, Ghent
  - University Hospital Leuven, Leuven

REFERENCES:
- See also: Related Info — http://www.uzgent.be